CLINICAL TRIAL: NCT03944798
Title: Surveillance AFter Extremity Tumor surgerY (SAFETY) International Randomized Controlled Trial
Brief Title: Surveillance AFter Extremity Tumor surgerY
Acronym: SAFETY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other); Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); American Academy of Orthopaedic Surgeons (Other); Musculoskeletal Tumor Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: GHRT02
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Soft Tissue Sarcoma; Lung Metastases
Keywords: Soft Tissue Sarcoma; Lung Metastases; Overall Survival; Surveillance; Randomized Controlled Trial; Patient Anxiety; Serious Adverse Events
MeSH Terms: conditions — Sarcoma | interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial superiority randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The local clinical team, site study personnel and participants cannot be blinded to the treatment allocation as the imaging modalities are visually distinguishable and these individuals will be required to arrange the booking of surveillance visits and imaging at their respective clinical site.
  The Central Adjudication Committee (CAC) will be blinded to surveillance frequency; however, because the imaging modalities are visually distinguishable, the CAC cannot be blinded to imaging modality. The data analysts will, however, remain blinded throughout the trial and all interpretation of study results will be conducted in a blinded manner. Since the primary outcome is objective, a lack of blinding of study personnel and patients, and the incomplete blinding of outcome assessors, introduces minimal threats to validity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Surveillance Arm I (Active Comparator): Clinical assessment and chest radiograph (CXR) every six months for two years
  Interventions: Other: Frequency: Every 6 Months; Other: Imaging Modality: Chest Radiograph (CXR)
- Surveillance Arm II (Experimental): Clinical assessment and CXR every three months for two years
  Interventions: Other: Frequency: Every 3 Months; Other: Imaging Modality: Chest Radiograph (CXR)
- Surveillance Arm III (Experimental): Clinical assessment and chest computed tomography (CT) every six months for two years
  Interventions: Other: Frequency: Every 6 Months; Other: Imaging Modality: Chest CT
- Surveillance Arm IV (Experimental): Clinical assessment and chest CT every three months for two years
  Interventions: Other: Frequency: Every 3 Months; Other: Imaging Modality: Chest CT

INTERVENTIONS:
Other: Frequency: Every 3 Months — every 3 months
  Arms: Surveillance Arm II; Surveillance Arm IV
Other: Frequency: Every 6 Months — every 6 months
  Arms: Surveillance Arm I; Surveillance Arm III
Other: Imaging Modality: Chest Radiograph (CXR) — Chest radiograph (CXR)
  Arms: Surveillance Arm I; Surveillance Arm II
Other: Imaging Modality: Chest CT — Chest computed tomography (CT)
  Arms: Surveillance Arm III; Surveillance Arm IV

SUMMARY:
Following treatment for a primary extremity sarcoma, patients remain at risk for the development of local and systemic disease recurrence. Metastasis (distant recurrence) to the lung is the most frequent single location of disease recurrence in sarcoma patients, occurring in almost half of all patients. Therefore, careful post-operative surveillance is an integral element of patient care. However, the detection of metastases does not necessarily affect long-term survival and may negatively impact quality of life. Surveillance strategies have not been well researched and have been identified as the top research priority in the extremity sarcoma field. Using a 2X2 factorial design to maximize efficiency and reduce overall trial costs, the SAFETY trial randomized 310 extremity soft-tissue sarcoma (STS) patients to determine the effect of surveillance strategy on overall patient survival after surgery for a STS of the extremity by comparing the effectiveness of both surveillance frequency (every 3 vs. every 6 months) and imaging modality (CT scans vs. chest radiographs).

DETAILED DESCRIPTION:
Post-treatment STS surveillance is an integral element of patient care. Although earlier detection of metastatic disease may improve long-term survival, no study has yet provided definitive evidence to support this assumption. A thorough systematic review of the literature has identified only a single limited randomized controlled trial (RCT) evaluating this clinical question, and surveys of sarcoma surgeons have determined that surgeons typically follow their patients based on the way in which they were trained. The orthopaedic oncology field has identified sarcoma surveillance strategy as the top research priority in the field. In order to fill the evidence gap in sarcoma surveillance, a large international RCT is required. The investigators, therefore, propose the Surveillance AFter Extremity Tumor surgerY (SAFETY) trial. In preparation for the SAFETY trial, the SAFETY investigators have completed the following preparatory work: A) establishment of a worldwide research collaborative group that spans 6 continents; B) collection of data from international sarcoma patients to determine their perceptions of sarcoma surveillance and their willingness to participate in a study in which randomization will determine their follow-up protocols; and C) the organization of a large Protocol Development Meeting with international and multidisciplinary participation, including sarcoma patient involvement, where critical aspects of the protocol were discussed and finalized.

The international, multi-center SAFETY trial will determine the effect of surveillance strategy on patient-important outcomes after surgery for a STS of the extremity by comparing the effectiveness of both surveillance frequency (every 3 vs. every 6 months) and imaging modality (CT scans vs. chest radiographs). Ultimately, the SAFETY trial will provide the necessary evidence to develop evidence-based surveillance guidelines, and is poised to have a significant impact on the post-operative care and outcomes of extremity STS patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years of age or older;
* The patient has been diagnosed with a primary extremity grade II or III soft-tissue sarcoma (STS);
* The patient has undergone surgical excision of the tumor with curative intent and with no evidence of gross residual disease based on the pathology report;
* The patient has completed all planned neoadjuvant or adjuvant radiation and / or chemotherapy, if applicable;
* The tumor size is greater than or equal to (≥) five centimeters according to the pathology report or based on the pre-treatment MRI if neoadjuvant radiation and / or chemotherapy are given; and
* The patient provides informed consent.

Exclusion Criteria:

* The patient has metastases at initial presentation based on the radiology report of the initial thoracic imaging†;
* The patient has recently undergone surgical excision of a local recurrence;
* The patient has been diagnosed with one of the special sub-types, myxoid / round cell liposarcoma or extra-skeletal Ewing's sarcoma*;
* The patient has been previously diagnosed with a genetic syndrome with an elevated risk of malignancy, such as Li-Freumeni Syndrome‡;
* The patient has been previously diagnosed with a co-morbid condition that has a life expectancy of less than (<) one year;
* The site-specific surveillance protocol for the patient's disease is not compatible with the study protocol (i.e., regular planned whole-body imaging with positron emission tomography [PET] scans);
* Likely problems, in the judgment of the investigator, with the patient maintaining follow-up (with the specific reasoning requiring approval of the Methods Center);
* The patient is currently enrolled in a study that does not permit co-enrolment; and
* The patient has already been enrolled in the SAFETY trial.

  * A second CT scan may be required to confirm that indeterminate nodules are false positives before the patient can be enrolled (provided that the second CT scan shows no evidence of metastatic disease);

    * Myxoid liposarcoma and extra-skeletal Ewing's sarcoma have different metastatic patterns, which necessitate different surveillance protocols;

      * Individuals with Li-Freumeni Syndrome, or other genetic syndromes with an elevated risk of malignancy, appear to be at an elevated risk for radiation-induced cancers, so the use of CT scans should be limited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Hierarchal Composite Outcome of Patient-Important Outcomes | 3 years post randomization
  The composite outcome consists of overall survival, serious adverse events, and patient-reported cancer-related anxiety

SECONDARY OUTCOMES:
Patient Anxiety | 3 years
  The PROMIS® Cancer-Anxiety instrument assesses self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). The PROMIS® Cancer-Anxiety instrument is a computer adaptive test. A minimum of 4 questions must be answered. One's responses will guide the system's choice of the next question. The test will continue until either the standard error drops below a specified level or the participant has answered the maximum number of 12 questions (whichever comes first). Each question has 5 response options ranging in value from 1 to 5. To find the raw score, sum the values of the response to each question. The lowest possible raw score is 4 and the highest is 60. The raw score will then be converted into a standardized T-score for each participant using the applicable conversion table. A higher T-score represents a higher degree of anxiety.
Patient Satisfaction | 3 years
  The PROMIS® Satisfaction with Social Roles & Activities instrument assesses satisfaction with performing one's usual social roles and activities (e.g., 'I am satisfied with my ability to participate in family activities'). This instrument is a computer adaptive test. A minimum of 4 questions must be answered. One's response will guide the system's choice of the next question. The test will continue until either the standard error drops below a specified level or the participant has answered the maximum number of 12 questions (whichever comes first). Each question has 5 response options ranging in value from 1 to 5. To find the raw score, sum the values of the response to each question. The lowest possible raw score is 4 and the highest possible raw score is 60. The raw score will then be converted into a standardized T-score for each participant using the applicable conversion table. A higher T-score represents a higher degree of satisfaction.
Patient Quality-of-Life | 3 years
  The validated EuroQol-5 Dimension 5-level (EQ-5D-5L) questionnaire measures generic health status and consists of 2 sections: the descriptive system and the Visual Analogue Scale (VAS). The descriptive system is comprised of 5 dimensions (mobility, self care, usual activities, pain / discomfort and anxiety / depression). Each question has 5 response options ranging in value from 1 to 5. To find the raw score, sum the values of the response to each question. The lowest possible raw score is 5 and the highest is 25. A lower raw score in the descriptive system represents fewer issues with each of the 5 domains. The VAS records a participant's self-rated health from 0 to 100 on a vertical VAS with endpoints labeled '100 - the best health you can imagine' and '0 - the worst health you can imagine'. The participant is asked to mark an 'X' on the scale and write the corresponding number, which is this section's raw score.
Local Recurrence-Free Survival | 3 years
  As measured by the length of time from the time of randomization that the participant survives with no detection of recurrent disease at the initial tumor site or operative field.
Metastasis-Free Survival | 3 years
  As measured by the length of time from the time of randomization that the participant survives with no detection of systemic disease recurrence at any anatomic location.
Treatment-Related Complications | 3 years
  Will include both chemotherapy-related complications, such as febrile neutropenia, fungal infections or sepsis, and thoracotomy-related complications, such as pneumothorax, or surgical site infections.
Net Healthcare Costs | 3 years
  Will include both the net costs of surveillance and costs incurred from metastasis treatment and metastasis treatment-related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ghert, MD, Principal Investigator — McMaster University
Locations (35):
- United States (16):
  - University of California Davis Medical Center, Sacramento, California
  - Hartford HealthCare, Hartford, Connecticut
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - UChicago Medicine, Chicago, Illinois
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - NYU Langone Orthopaedic Hospital/Perlmutter Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University Hospital, Portland, Oregon
  - Allegheny Health Network Research Institute, Monroeville, Pennsylvania
  - Texas Tech Health Sciences Center, El Paso, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Hospital Universitario Austral, Buenos Aires, Argentina
- St. Vincent's Hospital Melbourne, Fitzroy, Melbourne, Australia
- LKH - Universitätsklinikum Graz, Graz, Austria
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil
- Canada (7):
  - Nova Scotia Health, Halifax, Nova Scotia
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôtel Dieu du Quebec, Québec, Quebec
- Helios Klinikum Berlin, Berlin, Germany
- Centro Traumatologico Ortopedico Hospital, Turin, Italy
- University Malaya Kuala Lumpur, Kuala Lumpur, Malaysia
- Leiden University Medical Center, Leiden, Netherlands
- Centro Hospitalar e Universitario de Coimbra, Coimbra, Portugal
- Hospital Vall d'Hebron, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] SAFETY Investigators. The Surveillance After Extremity Tumor Surgery (SAFETY) trial: protocol for a pilot study to determine the feasibility of a multi-centre randomised controlled trial. BMJ Open. 2019 Sep 18;9(9):e029054. doi: 10.1136/bmjopen-2019-029054. PMID 31537562
- See also: Optimal surveillance strategies following curative surgery for extremity sarcoma: A systematic review of Randomized Control Trials [published in pre-print]. — http://osf.io/bnfsm/
- See also: Surveillance AFter Extremity Tumor surgerY (SAFETY): A Protocol for an International Randomized Controlled Trial [published in pre-print]. — http://osf.io/2wjyk/
- See also: The Surveillance After Extremity Tumor Surgery (SAFETY) Pilot International Multi-Center Randomized Controlled Trial — https://osf.io/preprints/osf/6h2um